CLINICAL TRIAL: NCT02475525
Title: The Role of an Arginine Enriched Oral Nutritional Supplement in the Prevention of Wound Complication in Patients Undergoing Lower Limb Revascularization
Brief Title: Oral Nutritional Supplement in Reducing Surgical Site Infections
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Recruitment difficulties
Sponsor: University of Limerick (Other)
Collaborators: UL Hospitals, Limerick (Unknown)
Responsible Party: Principal Investigator, Mary Clarke Moloney, Clinical Operations Manager, University of Limerick
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: ONS2015
Record Dates: First submitted 2015-06-08; First posted 2015-06-18 (Estimated); Last update posted 2018-05-04 (Actual); Status verified 2018-05

CONDITIONS: Peripheral Vascular Disease; Claudication
MeSH Terms: conditions — Peripheral Vascular Diseases; Intermittent Claudication

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arginine enriched oral nutritional supplement group (Experimental): Patients randomised to the oral nutritional supplement group will continue their normal diet. In addition, this group will commence taking oral nutritional supplement twice daily 5 days prior to surgery and continued for 4 weeks post surgery. Intake of nutritional drink will be suspended during their fasting period prior to surgery and will commence once surgery is completed and group are able to tolerate food post surgery. Wound examination will take place at 1 and at 4 weeks post surgery by the tissue viability nurse specialist who will be blinded to the treatment. Patient adherence to the study protocol with the nutritional supplement regimen will be recorded daily by the patient for four the four weeks the supplement is provided.
  Interventions: Dietary Supplement: Arginine enriched oral nutritional supplement
- Control (No Intervention): This group will continue on their normal diet before and after surgery. Normal diet will be suspended during their fasting period prior to surgery and will re commence once surgery is completed and group are able to tolerate food post surgery. Wound examination will take place at 1 and at 4 weeks post surgery by the tissue viability nurse specialist who will be blinded to the treatment.

INTERVENTIONS:
Dietary Supplement: Arginine enriched oral nutritional supplement — oral nutritional supplement containing arginine
  Other Names: CubitanTM
  Arms: Arginine enriched oral nutritional supplement group

SUMMARY:
The study aims to evaluate the efficacy of an arginine enriched oral nutritional supplement in the prevention of wound complications in the the wounds of patients post lower limb revascularization.

DETAILED DESCRIPTION:
Surgical incisions are associated with a number of possible complications. The reported incidence of surgical site infections at the groin after vascular procedures is between 3% and 30%. This incidence is up to five times higher than the expected incidence of infection in clean cases. Risk factors for postoperative surgical site infection in patients undergoing vascular surgery may include age, co-morbidities, use of prosthetic grafts and repeat operations.

A systematic review in 2011 concluded that arginine supplemented diets among perioperative patients were associated with a reduced rate of surgical infection and reduced overall length of hospital stay.

The study aims are to determine if taking an oral nutritional supplement reduces the rate of wound complications post lower limb revascularization.

ELIGIBILITY:
Inclusion Criteria:

* Patients scheduled for elective lower limb revascularization surgery
* patients aged >18 years.

Exclusion Criteria:

* Patients unable to provide informed consent,
* emergency cases,
* seriously ill patients/unconscious patients,
* chronic renal disease,
* known inflammatory bowel disease,
* known lactose intolerance and not using lactase,
* known galactosemia,
* pregnancy,
* cows milk allergy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2015-06 (Actual); Primary Completion 2016-12-01 (Actual); Study Completion 2017-02-01 (Actual)

PRIMARY OUTCOMES:
The number of incidents of wound infections in both groups of patients undergoing lower limb re vascularization. | 4 weeks

SECONDARY OUTCOMES:
Patient acceptability of the oral nutritional supplement. | 4 weeks
Duration of post operative hospital stay | 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Mary Clarke Moloney, Principal Investigator — University of Limerick; Paul Burke, Principal Investigator — UL Hospitals
Locations (1):
- University Hospital Limerick, Limerick, Ireland

IPD SHARING:
Plan to Share IPD: Undecided